CLINICAL TRIAL: NCT03200821
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of 250 µg G17DT or 1000 µg/m^2 Gemcitabine in Subjects With Advanced Pancreatic Cancer
Brief Title: An Open Label Study to Evaluate G17DT Compared to Gemcitabine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC3
Record Dates: First submitted 2017-05-30; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: A randomized, open, parallel group, active comparator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- G17DT (Experimental): 250 µg/0.2 mL administered by intramuscular injection at Weeks 0, 2 and 6. 125 µg booster administered at Week 24.
  Interventions: Biological: G17DT
- Gemcitabine (Active Comparator): 1000 µg/m^2 intravenously administered once weekly for seven weeks starting at Week 0 followed by one week of rest. After, treatments will occur in cycles of 3 weeks of treatment followed by one week of rest.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Biological: G17DT — 250 µg/0.2 mL administered by intramuscular injection at Weeks 0, 2 and 6. 125 µg booster administered at Week 24.
  Other Names: PAS, Polyclonal Antibody Stimulator
  Arms: G17DT
Drug: Gemcitabine — 1000 µg/m^2 intravenously administered once weekly for seven weeks starting at Week 0 followed by one week of rest. After, treatments will occur in cycles of 3 weeks of treatment followed by one week of rest.
  Other Names: Gemzar
  Arms: Gemcitabine

SUMMARY:
In this study 250 µg of G17DT was administered at Weeks 0, 2 and 6 in order to demonstrate non inferiority compared to gemcitabine in prolonging survival in advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of pancreatic adenocarcinoma, confirmed by histology or cytology, in patients not suitable for pancreatic tumor resection with curative intent.
* A diagnosis of recurrent pancreatic adenocarcinoma (previously confirmed by histology or cytology) in patients who have had a primary tumor resection.
* Male or female patients over 18 years of age.
* Laboratory values within the following ranges at screening:

Serum creatinine < 1.25 times upper limit of normal (ULN) Haemoglobin > 9.5 g/dL White blood cell (WBC) count > 3.5 x 109/L Platelets > 100 x 109/L Total bilirubin < 2.0 times ULN Aspartate transaminase (AST, SGOT) < 3 times ULN

* A life expectancy of at least 2 months.
* A negative pregnancy test at the screening visit (females of childbearing potential only).
* Signed written informed consent.

Exclusion Criteria:

* History of other malignant disease (except basal cell carcinoma or in situ carcinoma of the uterine cervix).
* Previous cytotoxic chemotherapy (including gemcitabine).
* Previous radiotherapy within 30 days of baseline.
* Use of systemic (oral or injected) immunosuppressants, including corticosteroids, within 30 days prior to the baseline visit. Inhaled corticosteroids for chronic obstructive pulmonary disease or asthma were permitted.
* Females of child bearing potential who are pregnant, lactating, or who are planning to become pregnant during the period of the study.
* Participation in another study involving an investigational drug within 90 days of baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2000-08-14 (Actual); Primary Completion 2001-09-24 (Actual); Study Completion 2002-09-19 (Actual)

PRIMARY OUTCOMES:
Survival | Baseline (Week 0) up to Week 52 or death.
  Survival in days measured starting at Baseline

SECONDARY OUTCOMES:
Tumor Response | Weeks 0, 12, 24, 36 and 52
  The proportion of patients having an objective tumor response using Computed Tomography (CT) and the Response Evaluation Criteria In Solid Tumors (RECIST).
  (RECIST) guidelines
Quality of Life | Weeks 0, 6, 12, 24, 36 and 52
  Quality of life measured using Cancer Quality of Life Questionnaire EORTC-QLQC30 questionnaire
Quality of Life | Weeks 0, 6, 12, 24, 36 and 52
  Quality of life measured using and the EORTC QLQ-PAN26 questionnaire
Karnofsky Performance Status | Week 0 to Week 52
  Functional impairment assessment using the Karnofsky Performance Scale Index
Gastrin-17 Antibodies | Weeks 0, 6, 12, 24, 36 and 52
  Antibody assessment to determine serum levels of Gastrin -17 antibodies

IPD SHARING:
Plan to Share IPD: No